CLINICAL TRIAL: NCT04207463
Title: A Phase II, Open, Single-arm, Multi-cohort, Multicenter Study of Anlotinib and AK105 Injection in Subjects With Gastrointestinal Tumors, Urinary System Tumors, Neuroendocrine Tumors
Brief Title: A Study of Anlotinib and AK105 Injection in Subjects With Gastrointestinal Tumors, Urinary System Tumors, Neuroendocrine Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-AK105-II-02
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Gastrointestinal Tumors, Urinary System Tumors, Neuroendocrine Tumors
MeSH Terms: conditions — Digestive System Neoplasms; Neuroendocrine Tumors | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib and AK105 injection (Experimental): AK105 200mg intravenously (IV) on day 1 of each 21-day cycle plus Anlotinib capsules given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: AK105; Drug: Anlotinib

INTERVENTIONS:
Drug: AK105 — AK105 is a humanized monoclonal antibody that specifically binds to PD-1. AK105 has a typical antibody structure and is composed of two lgG1 subtype heavy chains and two kappa subtypes light chains covalently linked by disulfide bonds.
Drug: Anlotinib — a multi-target receptor tyrosine kinase inhibitor

SUMMARY:
AK105 is a humanized monoclonal antibody that specially binds to PD-1. Anlotinib is a small molecule tyrosine kinase inhibitor. Based on the mechanism study, tumor vascular abnormalities promote tissue hypoxia and increase lactic acid, thereby activating immunosuppression and inhibiting T cell function. Anti-angiogenic drugs enhance the infiltration of effector immune cells by inducing normalization of blood vessels and reducing immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* 1. Cohort 1：Histopathologically confirmed metastatic or inoperable cholangiocarcinoma failed with first-line or above chemotherapy.

Cohort 2： Histopathologically confirmed recurrent or metastatic colorectal cancer that is not suitable for surgery with MSI-H or dMMR.

Cohort 3： Histopathologically confirmed metastatic or recurrent gastric or gastroesophageal junction (GEJ) adenocarcinoma.

Cohort 4：Histopathologically confirmed local progression or metastatic urothelial carcinoma that is not suitable for surgery.

Cohort 5：Low- and medium-grade (G1 or G2) late gastrointestinal pancreatic neuroendocrine tumor (NET) subjects diagnosed by pathology." 2.18 years and older; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; Life expectancy ≥ 3 months.

3.At least one measurable lesion. 4.The main organs function are normally. 5. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

6. Understood and signed an informed consent form.

Exclusion Criteria:

* 1.Has used anti-angiogenic drugs such as bevacizumab, erlotinib, apatinib, sorafenib, sunitinib, and endothelium or against PD-1, PD-L1 and other related immunotherapeutic drugs.

  2. HER2 positive in cohort 3. 3. Has received chemotherapy, radiotherapy or other treatments within 4 weeks prior to the first dose.

  4.Has brain metastases with symptoms or symptoms control for less than 2 months.

  5.Has diagnosed and/or treated additional malignancy within 5 years prior to the first dose.

  6.Has multiple factors affecting oral medication. 7.Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.

  8.Has unrelieved spinal cord compression. 9.Imaging shows that tumors invade large blood vessels. 10.Has hemoptysis within 1 month prior to the first dose and maximum daily hemoptysis ≥2.5 mL.

  11.Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1.

  12.Has received surgery, or unhealed wounds within 4 weeks before the first dose.

  13. Has artery/venous thrombosis prior to the first dose within 6 months. 14. Has drug abuse history that unable to abstain from or mental disorders 15. Has any serious and / or uncontrolled disease. 16. Has received vaccination or attenuated vaccine within 4 weeks prior to the first dose.

  17.Hypersensitivity to recombinant humanized anti-PD-1 monoclonal or its components.

  18. Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first dose.

  19.Diagnosed as immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose >10 mg/day of prednisone or other therapeutic hormones) and continued to be used for 2 weeks prior to the first dose 20. Has participated in other anticancer drug clinical trials within 4 weeks. 21. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Disease control rate（DCR） | up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 96 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.
Progression-free survival (PFS) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) | up to 120 weeks
  OS defined as the time from the first dose to death from any cause. Subjects who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Harbin Medical University Cancer Hospital, Harbin, Jilin
  - Jinan Central Hospital, Jinan, Shandong
  - Shanxi Provincial Cancer Hospital, Xi’an, Shanxi